CLINICAL TRIAL: NCT04338243
Title: Open Label, Multicenter Phase Ib / II Study of Glumetinib Combined With Osimertinib in the Treatment of Relapsed and Metastatic Non-small Cell Lung Cancer Patients Who Failed to Receive EGFR Inhibitors
Brief Title: Glumetinib Combined With Osimertinib in the Treatment of Relapsed and Metastatic Non-small Cell Lung Cancer Patients Who Failed to Receive EGFR Inhibitors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCC244-203
Record Dates: First submitted 2020-03-29; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Negative T790M Mutation and Met Amplification
Keywords: MET amplification， T790
MeSH Terms: interventions — glumetinib

STUDY DESIGN:
Intervention Model Description: Phase Ib: Glumetinib 300mg Combined With Osimertinib 80mg, Qd ,oral
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glumetinib+Osimertinib (Experimental): The investigational product Glumetinib will be orally administrated when fasting at dose level of 300mg QD and Osimertinib will be orally administrated when fasting at dose level of 80mg QD
  Interventions: Drug: Glumetinib

INTERVENTIONS:
Drug: Glumetinib — Phase Ib is a dose escalation study, the initial dose of Glumetinib is 300mg, then will be escalated to 400mg，according to the result of Phase Ib， will confirm the RP2D

SUMMARY:
To explore the safety and efficacy of Glumetinib combined with Osimertinib in the treatment of relapsed and metastatic non-small cell lung cancer (NSCLC) with failed first-generation or second-generation EGFR inhibitors, negative T790M mutation and met amplification.

DETAILED DESCRIPTION:
To explore the safety and efficacy of Glumetinib combined with Osimertinib in the treatment of relapsed and metastatic non-small cell lung cancer (NSCLC) with failed first-generation or second-generation EGFR inhibitors, negative T790M mutation and met amplification.

ELIGIBILITY:
Inclusion Criteria:

* Can fully understand and sign informed consent form(ICF) voluntarily Male and female patients 18-80 (inclusive) years of age
* Stage: IIIb/IIIc/IV (AJCC version 8)
* ECOG Performance Status (PS): 0-1
* At least one measurable lesion as per RECIST 1.1

Exclusion Criteria:

* Subjects with characterizedALK or ROS1 activating mutations that predict sensitivity to anti-ALK-therapy or anti-ROS1-therapy; T790 mutations is uknown or positive
* Patients who have symptomatic CNS metastasis which is neurologically unstable or those who have CNS disease requiring increase in the dose of steroid. (Note: Patients with controlled CNS metastasis can participate in the trial. Before entering the study, patients should have finished radiotherapy, or have received operation for CNS tumor metastasis at least two weeks before. Patients' neurological function must be in a stable state; no new neurological deficit is found during clinical examination and no new problem is found during CNS imaging examinations. If patients need to use steroids to treat CNS metastasis, the therapeutic dose of steroid should be stable for ≥3 months at least two weeks prior to entering the study.)
* Prior exposure to MET-directed or third generation EGFR inhibitors therapy Anticancer therapy (including chemotherapy, targeted therapy, biotherapy, hormone therapy or other investigational agents) within 4 weeks or 5 times of half-lives (whichever is shorter) prior to the first dose of the study drug or who have not recovered from the side effect of such therapy
* Major surgery or had significant traumatic injury within 28 days prior to the first dose of the investigational product

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective response rate) | through study completion, an average of 1 year
  the sum ratio of partial response and complete response(determined by an Independent Radiology Review Committee (IRRC) according to RECIST Version 1.1)

SECONDARY OUTCOMES:
ORR(Objective response rate, assessed as per investigators) | through study completion, an average of 1 year
  the sum ratio of partial response and complete response(assessed as per investigators)
DOR(Duration of response) | The time from the date of first documented partial response or complete response to progressive disease or death, an average of 6 months
  The time from the partial response and complete response of patient to patient progressive disease or death
OS(Overall survival) | Through study completion, an average of 1 year
  The time from the patient first dose to death

CONTACTS AND LOCATIONS:
Overall Officials: Yongqian Shu, Doctor, Principal Investigator — Jiangsu Province People's Hospital; Dingzhi Huang, Doctor, Principal Investigator — Tianjin Cancer Hospital; Yiping Zhang, Doctor, Principal Investigator — Zhejiang Province Cancer Hospital; Jianying Zhou, Doctor, Principal Investigator — Zhejiang University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided